CLINICAL TRIAL: NCT00635440
Title: The Effect of Neuromuscular Electrical Stimulation on Muscle Metabolism of Major Abdominal Surgical Patients
Brief Title: Randomized, Controlled Study to Investigate the Effect of Neuromuscular Electrical Stimulation (NMES) on Muscle Metabolism of Abdominal Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Department of Surgery, Social Medical Centre South, Vienna, Austria (Unknown); Institute for Pathology and Microbiology, Social Medical Centre South, Vienna, Austria (Unknown)
Responsible Party: Institute of Physical Medicine and Rehabilitation, Social Medical Centre South, Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Muscle-2446
Record Dates: First submitted 2008-02-25; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Muscular Atrophy
Keywords: skeletal muscle; ubiquitin; proteasome; IGF-1; MGF; protein catabolism; neuromuscular electrical stimulation; Investigate effect of NMES on muscle metabolism of catabolic patients
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Device: neuromuscular electrical stimulation: Cefar-Sport (CefarCompex Scandinavia AB)
- B (Sham Comparator)
  Interventions: Device: neuromuscular electrical stimulation: Cefar-Sport (CefarCompex Scandinavia AB)

INTERVENTIONS:
Device: neuromuscular electrical stimulation: Cefar-Sport (CefarCompex Scandinavia AB) — Electrical stimuli of 50 Hz (pulse width 0.25ms, 8 sec on, 4 sec off) were applied daily for 30 min, for 4 days, starting on the first postoperative day.The amplitude of the electrical stimuli in the stimulated leg was adjusted to ensure maximum tolerable muscle contraction.
  Arms: A
Device: neuromuscular electrical stimulation: Cefar-Sport (CefarCompex Scandinavia AB) — Electrical stimuli of 50 Hz (pulse width 0.25ms, 8 sec on, 4 sec off) were applied daily for 30 min, for 4 days, starting on the first postoperative day. Current was increased until the patient could feel a tingling sensation but no muscle contraction was visible or palpable.
  Arms: B

SUMMARY:
Skeletal muscle atrophy is associated with catabolic conditions such as major surgical interventions and leads to reduced muscle strength, increased clinical complications and prolonged convalescence. Several studies revealed immobilisation as a major stimulus for muscle wasting in severely ill patients. This study investigates the potency of neuromuscular electrical stimulation on skeletal muscle growth factors and degradation processes in major abdominal surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* intended for major abdominal surgery
* more than 18 years old

Exclusion Criteria:

* neuromuscular diseases
* immobility before surgery
* arterial occlusive disease Fontaine stadium IV
* clinical or laboratory signs of inflammation or sepsis
* cachexia
* diseases of the musculoskeletal systems contraindicating electrical stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-12

PRIMARY OUTCOMES:
mRNA level of IGF-1Ea

SECONDARY OUTCOMES:
mRNA level of MGF, total RNA content, total protein content, ubiquitin conjugated proteins, proteasome activity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quittan, PhD, MD, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Social Medical Centre South
Locations (1):
- Institute of Physical Medicine and Rehabilitation, Social Medical Centre South, Vienna, Vienna, Austria

REFERENCES:
- [Background] Roth E, Valentini L, Holzenbein T, Winkler S, Sautner T, Hortnagl H, Karner J. Acute effects of insulin-like growth factor I on inter-organ amino acid flux in protein-catabolic dogs. Biochem J. 1993 Dec 15;296 ( Pt 3)(Pt 3):765-9. doi: 10.1042/bj2960765. PMID 8280075
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Biolo G, Ciocchi B, Lebenstedt M, Barazzoni R, Zanetti M, Platen P, Heer M, Guarnieri G. Short-term bed rest impairs amino acid-induced protein anabolism in humans. J Physiol. 2004 Jul 15;558(Pt 2):381-8. doi: 10.1113/jphysiol.2004.066365. Epub 2004 May 6. PMID 15131238
- [Background] DeVol DL, Rotwein P, Sadow JL, Novakofski J, Bechtel PJ. Activation of insulin-like growth factor gene expression during work-induced skeletal muscle growth. Am J Physiol. 1990 Jul;259(1 Pt 1):E89-95. doi: 10.1152/ajpendo.1990.259.1.E89. PMID 2372054
- [Background] Hameed M, Orrell RW, Cobbold M, Goldspink G, Harridge SD. Expression of IGF-I splice variants in young and old human skeletal muscle after high resistance exercise. J Physiol. 2003 Feb 15;547(Pt 1):247-54. doi: 10.1113/jphysiol.2002.032136. Epub 2002 Dec 20. PMID 12562960
- [Background] Bodine SC, Latres E, Baumhueter S, Lai VK, Nunez L, Clarke BA, Poueymirou WT, Panaro FJ, Na E, Dharmarajan K, Pan ZQ, Valenzuela DM, DeChiara TM, Stitt TN, Yancopoulos GD, Glass DJ. Identification of ubiquitin ligases required for skeletal muscle atrophy. Science. 2001 Nov 23;294(5547):1704-8. doi: 10.1126/science.1065874. Epub 2001 Oct 25. PMID 11679633
- [Background] Quittan M, Wiesinger GF, Sturm B, Puig S, Mayr W, Sochor A, Paternostro T, Resch KL, Pacher R, Fialka-Moser V. Improvement of thigh muscles by neuromuscular electrical stimulation in patients with refractory heart failure: a single-blind, randomized, controlled trial. Am J Phys Med Rehabil. 2001 Mar;80(3):206-14; quiz 215-6, 224. doi: 10.1097/00002060-200103000-00011. PMID 11237275
- [Derived] Strasser EM, Stattner S, Karner J, Klimpfinger M, Freynhofer M, Zaller V, Graf A, Wessner B, Bachl N, Roth E, Quittan M. Neuromuscular electrical stimulation reduces skeletal muscle protein degradation and stimulates insulin-like growth factors in an age- and current-dependent manner: a randomized, controlled clinical trial in major abdominal surgical patients. Ann Surg. 2009 May;249(5):738-43. doi: 10.1097/SLA.0b013e3181a38e71. PMID 19387331